CLINICAL TRIAL: NCT02719054
Title: Effect of Community Based Depression Management and Psychosocial Stimulation Intervention on Maternal Mental Health and Child Development: A Randomized Controlled Trial
Brief Title: Effect of Community Based Depression Management and Child Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bangor University (Other); Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-13066
Record Dates: First submitted 2016-03-02; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Maternal Depressive Symptom and Child Development
Keywords: Depression; Child Development; Stimulation; CBT; Bangladesh
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stimulation (Experimental): Cognitive behavioral therapy for mother and play stimulation for children aged 6 to 12 months
  Interventions: Behavioral: Cognitive behavioral therapy: Alter of negative thinking, positive thinking and social support and psychosocial stimulation: play stimulation and parenting
- Mother child dyad (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy: Alter of negative thinking, positive thinking and social support and psychosocial stimulation: play stimulation and parenting — A:Cognitive Behavioral Therapy specifically focused on "changing thinking style toward positive" and not associated with any medication. CBT found to be effective in managing or treating not only depression, also a variety of other conditions-e.g. mood, personality, stress, eating habit, tic etc.
  B: Psycho social stimulation will follow a set of culturally appropriate, semi-structured, child's age appropriate curriculum.
  Other Names: CBT & PS
  Arms: stimulation

SUMMARY:
Investments in Early childhood Development (ECD) programs produce higher economic return through maximizing human potential. In developing countries over 200 million children do not reach their developmental potential. Early nutritional support and psycho social stimulation are essential for optimum development of children. Mothers are usually the key providers of childcare.

Depression is reported as a leading cause of disease burden for women and maternal mental health is identified as one of the major predictors of child development.

In Bangladesh, almost 60% children are at risk of poor development due to high prevalence of Low Birth Weight (22%), under nutrition (41%), poverty, and sub-optimal stimulation. About one third of Bangladeshi mothers suffer from depression. Early stimulation interventions in Bangladesh have showed moderate improvements to children's development. This indicates that there are still some gaps in the pathway to delivery. So, it is crucially important to address maternal mental health along with any Early Childhood Development intervention at community level to get bigger impact.

In Bangladesh mothers with sub clinical depressive symptoms often do not seek treatment due to the stigma attached to it. Depressed mothers who do not receive treatment often fail to provide sufficient stimulation and care for their children and in turn compromise benefits of early stimulation programs. Rahman and colleagues (2008) tested an innovative model of community-based depression management using Cognitive Behavioral Therapy in Pakistan and reported improvement in maternal depression 6 months postpartum.

The study plans to combine the above treatment of depression with an evidenced-based Early Childhood Development program to achieve maximum benefits on reducing maternal depressive symptoms as well as improving children's overall development.

DETAILED DESCRIPTION:
Present study proposes to conduct the study in rural areas covered by community clinic (CC) services and will use their community based staff to deliver the intervention. Each Community Clinic is established at grass root level providing one stop service center for Primary Health Care for approx. 6000 population. There are over 12000 Community Clinics operating in Bangladesh. We chose this population as almost 75% of people live in rural areas and they will form a representative sample for scaling in future. There will be 2 groups in the study i) Intervention group (Cognitive Behavioral Therapy + play stimulation) and ii) control group (with none)..

Previous studies reported moderate benefit with both home and center based psycho social stimulation program in Bangladesh. However in most parts we found low self esteem among the mothers that required quite effort to bring them into the task. So it is assumed that the proposed community based Cognitive Behavioral Therapy model (Rahman et al 2008) for management of depressive symptoms, will be a unique sustainable approach to get maximize effect psycho social stimulation intervention. The study aimed to deliver the intervention using government health infrastructure. The study will evaluate the workload of existing 2 staff -Health Assistant (HA) and Family Welfare Assistant (FWA) at each Community Clinic who regularly go for home visits and will train them for intervention. The study may need to train one additional person from the same community to assist Health Assistant or Family Welfare Assistant in delivering the intervention. The overall success of the project will be able to come up with a model that can be used by other Community Clinics to take it to scale.

After selection of study sites under 30 Community Clinics, randomization will be done. The study will do several small group discussions with mothers living in those communities to know about their lifestyle, local terminologies of depressive symptoms, view about depressive symptoms, child rearing practices and coping strategies. Then Health Assistants and Family Welfare Assistants of 15 intervention Community Clinics will be identified and will receive training in batches. In next step, after taking consent, screening will be conducted in the community among mothers of 9-12 months old children by trained psychologists. Considering the Community Clinics as a center, data collectors will start screening from center to periphery in the community until we get 10 mothers with depressive symptoms. Mothers, who will fulfill the study enrollment criteria, will be offered to join the study and will be invited to the test center for baseline assessment (of mother-child dyad). We will set up temporary test centers in villages under each Community Clinic, using a space in Community Clinics (provided there is available space) or rooms in schools or convenient rented rooms in residence of local people. Two teams of testers and interviewers will be rotated from one Community Clinic to another after completing screening and baseline psychological assessments in areas under that Community Clinic which on average would take 2-3 days. It is expected that the baseline assessment will be covered by 2 months. Soon after baseline assessment in one Community Clinic, intervention in villages under that Community Clinic will be started by the trained Health Assistant/Family Welfare Assistant assigned to that Community Clinic. In the middle of the study, the study will conduct in-depth interview on two mothers under each Community Clinic to know about mothers' perception and comments about the intervention for further modification of the program. The study will also conduct small group discussions with the Health Assistant and Family Welfare Assistant about the intervention during monthly meetings with them- to know their views about the program. After 12 months intervention, final assessment will be done following the same procedure"

ELIGIBILITY:
Inclusion Criteria:

* Mother with depressive symptom( EPDS ≥10) with child aged 6 to 12 months

Exclusion Criteria:

* Mother with known severe chronic diseases
* Children with known severe chronic diseases

Ages: 6 Months to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Child's cognitive, motor and language and behavioral assessment( developmental out come) | At base line and change of develomental outcome after one year of intervention at end line
  Child's cognitive, motor and language assessment using Bayley-III and behavioral assessment during test using Wolke's Behavior Rating Scale. Wolke,s Behavior Rating scale is used through observation during Bayley test. Bayley test includes cognitive, motor and language development. All outcomes will have quantitative scores and results will be made adding the scores.
Depressive symptoms | At base line and change of depressive symptomatic outcome after one year of intervention at end line
  Depression Scores using Edinburgh Postpartum Depression Scale (EPDS) at baseline (during screening at home) and at the end. Result will be made adding score of each questions.
Mother's self esteem | At base line and change of state of mother's self esteem after one year of intervention at end line
  This will be assessed using adapted version of the Rosenberg Self Esteem Scale, the most widely used measure of self esteem for research purposes. It has been used previously in Bangladesh by our team as a valid instrument.
Family Care Indicators | At base line and change of Family Care Indicator after one year of intervention at end line
  This will be used to measure quality of stimulation the child received at home. FCI has been used in Bangladesh previously and showed good reliabilities
Child care knowledge and practices | At base line and change of care giver's child care knowledge and practice after one year of intervention at end line
  A modified questionnaire based on our previous studies (Hamadani et al. 2006; Nahar et al. 2012) will be given to mothers to assess child care practices.

SECONDARY OUTCOMES:
Children's height | At base line and change of children's height after one year of intervention at end line.
  Children's height at baseline and at the end in test centre. Both the children of control and intervention group may have some medical problems. So as the problems are for the both groups the study results will not be much varied.
Children's weight | At base line and change of children's weight after one year of intervention at end line.
  Children's weight at baseline and at the end in test centre. Both the children of control and intervention group may have some medical problems. So as the problems are for the both groups the study results will not be much varied.
Children's Mid Upper Arm Circumference (MUAC) | At base line and change of children's weight after one year of intervention at end line.
  Children's Mid Upper Arm Circumference (MUAC) at baseline and at the end in test center. Both the children of control and intervention group may have some medical problems. So as the problems are for the both groups the study results will not be much varied.
Children's Occipital Frontal Circumference | At base line and change of children's Occipital Frontal Circumference after one year of intervention at end line.
  Children's Occipital Frontal Circumference at baseline and at the end in test center. Both the children of control and intervention group may have some medical problems. So as the problems are for the both groups the study results will not be much varied.
Mother's height | At base line and change of mother's height after one year of intervention at end line.
  Mother's height at baseline and at the end in test center. Both the mothers of control and intervention group may have some medical problems. So as the problems are for the both groups the study results will not be much varied.
Mother's height | At base line and change of mother's weight after one year of intervention at end line.
  Mother's weight at baseline and at the end in test center. Both the mothers of control and intervention group may have some medical problems. So as the problems are for the both groups the study results will not be much varied.

IPD SHARING:
Plan to Share IPD: Yes
We will share data with our collaborators

REFERENCES:
- [Result] Black MM, Baqui AH, Zaman K, McNary SW, Le K, Arifeen SE, Hamadani JD, Parveen M, Yunus M, Black RE. Depressive symptoms among rural Bangladeshi mothers: implications for infant development. J Child Psychol Psychiatry. 2007 Aug;48(8):764-72. doi: 10.1111/j.1469-7610.2007.01752.x. PMID 17683448
- [Result] Engle PL, Fernald LC, Alderman H, Behrman J, O'Gara C, Yousafzai A, de Mello MC, Hidrobo M, Ulkuer N, Ertem I, Iltus S; Global Child Development Steering Group. Strategies for reducing inequalities and improving developmental outcomes for young children in low-income and middle-income countries. Lancet. 2011 Oct 8;378(9799):1339-53. doi: 10.1016/S0140-6736(11)60889-1. Epub 2011 Sep 22. PMID 21944378
- [Result] Gausia K, Hamadani JD, Islam MM, Ali M, Algin S, Yunus M, Fisher C, Oosthuizen J. Bangla translation, adaptation and piloting of Edinburgh Postnatal Depression Scale. Bangladesh Med Res Counc Bull. 2007 Dec;33(3):81-7. doi: 10.3329/bmrcb.v33i3.1138. PMID 18783062
- [Result] Grantham-McGregor SM, Lira PI, Ashworth A, Morris SS, Assuncao AM. The development of low birth weight term infants and the effects of the environment in northeast Brazil. J Pediatr. 1998 Apr;132(4):661-6. doi: 10.1016/s0022-3476(98)70357-9. PMID 9580767
- [Result] Grantham-McGregor S; International Child Development Committee. Early child development in developing countries. Lancet. 2007 Mar 10;369(9564):824. doi: 10.1016/S0140-6736(07)60404-8. No abstract available. PMID 17350449
- [Result] Hamadani JD, Fuchs GJ, Osendarp SJ, Khatun F, Huda SN, Grantham-McGregor SM. Randomized controlled trial of the effect of zinc supplementation on the mental development of Bangladeshi infants. Am J Clin Nutr. 2001 Sep;74(3):381-6. doi: 10.1093/ajcn/74.3.381. PMID 11522564
- [Result] Hamadani JD, Fuchs GJ, Osendarp SJ, Huda SN, Grantham-McGregor SM. Zinc supplementation during pregnancy and effects on mental development and behaviour of infants: a follow-up study. Lancet. 2002 Jul 27;360(9329):290-4. doi: 10.1016/S0140-6736(02)09551-X. PMID 12147372
- [Result] Hamadani JD, Huda SN, Khatun F, Grantham-McGregor SM. Psychosocial stimulation improves the development of undernourished children in rural Bangladesh. J Nutr. 2006 Oct;136(10):2645-52. doi: 10.1093/jn/136.10.2645. PMID 16988140
- [Result] Hamadani JD, Tofail F, Hilaly A, Huda SN, Engle P, Grantham-McGregor SM. Use of family care indicators and their relationship with child development in Bangladesh. J Health Popul Nutr. 2010 Feb;28(1):23-33. doi: 10.3329/jhpn.v28i1.4520. PMID 20214083
- [Result] Idjradinata P, Pollitt E. Reversal of developmental delays in iron-deficient anaemic infants treated with iron. Lancet. 1993 Jan 2;341(8836):1-4. doi: 10.1016/0140-6736(93)92477-b. PMID 7678046
- [Result] Karasz A. Cultural differences in conceptual models of depression. Soc Sci Med. 2005 Apr;60(7):1625-35. doi: 10.1016/j.socscimed.2004.08.011. PMID 15652693
- [Result] Khan MM, Reza H. The pattern of suicide in Pakistan. Crisis. 2000;21(1):31-5. doi: 10.1027//0227-5910.21.1.31. PMID 10793469
- [Result] Khan MM, Reza H. Gender differences in nonfatal suicidal behavior in Pakistan: significance of sociocultural factors. Suicide Life Threat Behav. 1998 Spring;28(1):62-8. PMID 9560167
- [Result] Kumar V. Poisoning deaths in married women. J Clin Forensic Med. 2004 Feb;11(1):2-5. doi: 10.1016/j.jcfm.2003.10.010. PMID 15261005
- [Result] Lawrence V, Murray J, Banerjee S, Turner S, Sangha K, Byng R, Bhugra D, Huxley P, Tylee A, Macdonald A. Concepts and causation of depression: a cross-cultural study of the beliefs of older adults. Gerontologist. 2006 Feb;46(1):23-32. doi: 10.1093/geront/46.1.23. PMID 16452281
- [Result] Lind T, Lonnerdal B, Stenlund H, Gamayanti IL, Ismail D, Seswandhana R, Persson LA. A community-based randomized controlled trial of iron and zinc supplementation in Indonesian infants: effects on growth and development. Am J Clin Nutr. 2004 Sep;80(3):729-36. doi: 10.1093/ajcn/80.3.729. PMID 15321815
- [Result] Lovejoy MC, Graczyk PA, O'Hare E, Neuman G. Maternal depression and parenting behavior: a meta-analytic review. Clin Psychol Rev. 2000 Aug;20(5):561-92. doi: 10.1016/s0272-7358(98)00100-7. PMID 10860167
- [Result] Murray L, Cooper P. Effects of postnatal depression on infant development. Arch Dis Child. 1997 Aug;77(2):99-101. doi: 10.1136/adc.77.2.99. No abstract available. PMID 9301345
- [Result] Nahar B, Hamadani JD, Ahmed T, Tofail F, Rahman A, Huda SN, Grantham-McGregor SM. Effects of psychosocial stimulation on growth and development of severely malnourished children in a nutrition unit in Bangladesh. Eur J Clin Nutr. 2009 Jun;63(6):725-31. doi: 10.1038/ejcn.2008.44. Epub 2008 Sep 3. PMID 18772893
- [Result] Nahar B, Hossain MI, Hamadani JD, Ahmed T, Huda SN, Grantham-McGregor SM, Persson LA. Effects of a community-based approach of food and psychosocial stimulation on growth and development of severely malnourished children in Bangladesh: a randomised trial. Eur J Clin Nutr. 2012 Jun;66(6):701-9. doi: 10.1038/ejcn.2012.13. Epub 2012 Feb 22. PMID 22353925
- [Result] Nahar B, Hossain MI, Hamadani JD, Ahmed T, Grantham-McGregor S, Persson LA. Effects of psychosocial stimulation on improving home environment and child-rearing practices: results from a community-based trial among severely malnourished children in Bangladesh. BMC Public Health. 2012 Aug 7;12:622. doi: 10.1186/1471-2458-12-622. PMID 22871096
- [Result] Nasreen HE, Kabir ZN, Forsell Y, Edhborg M. Prevalence and associated factors of depressive and anxiety symptoms during pregnancy: a population based study in rural Bangladesh. BMC Womens Health. 2011 Jun 2;11:22. doi: 10.1186/1472-6874-11-22. PMID 21635722
- [Result] Najman JM, Andersen MJ, Bor W, O'Callaghan MJ, Williams GM. Postnatal depression-myth and reality: maternal depression before and after the birth of a child. Soc Psychiatry Psychiatr Epidemiol. 2000 Jan;35(1):19-27. doi: 10.1007/s001270050004. PMID 10741532
- [Result] Patel V, Araya R, Bolton P. Treating depression in the developing world. Trop Med Int Health. 2004 May;9(5):539-41. doi: 10.1111/j.1365-3156.2004.01243.x. No abstract available. PMID 15117296
- [Result] Patel V, Rahman A, Jacob KS, Hughes M. Effect of maternal mental health on infant growth in low income countries: new evidence from South Asia. BMJ. 2004 Apr 3;328(7443):820-3. doi: 10.1136/bmj.328.7443.820. PMID 15070641
- [Result] Pollitt E, Saco-Pollitt C, Jahari A, Husaini MA, Huang J. Effects of an energy and micronutrient supplement on mental development and behavior under natural conditions in undernourished children in Indonesia. Eur J Clin Nutr. 2000 May;54 Suppl 2:S80-90. doi: 10.1038/sj.ejcn.1601009. PMID 10902991
- [Result] Rahman A, Iqbal Z, Harrington R. Life events, social support and depression in childbirth: perspectives from a rural community in the developing world. Psychol Med. 2003 Oct;33(7):1161-7. doi: 10.1017/s0033291703008286. PMID 14580070
- [Result] Rahman A, Malik A, Sikander S, Roberts C, Creed F. Cognitive behaviour therapy-based intervention by community health workers for mothers with depression and their infants in rural Pakistan: a cluster-randomised controlled trial. Lancet. 2008 Sep 13;372(9642):902-9. doi: 10.1016/S0140-6736(08)61400-2. PMID 18790313
- [Result] Raj A, Silverman JG. Intimate partner violence against South Asian women in greater Boston. J Am Med Womens Assoc (1972). 2002 Spring;57(2):111-4. PMID 11991419
- [Result] Schellenberg JA, Victora CG, Mushi A, de Savigny D, Schellenberg D, Mshinda H, Bryce J; Tanzania Integrated Management of Childhood Illness MCE Baseline Household Survey Study Group. Inequities among the very poor: health care for children in rural southern Tanzania. Lancet. 2003 Feb 15;361(9357):561-6. doi: 10.1016/S0140-6736(03)12515-9. PMID 12598141
- [Result] Segre LS, Stasik SM, O'Hara MW, Arndt S. Listening visits: an evaluation of the effectiveness and acceptability of a home-based depression treatment. Psychother Res. 2010 Nov;20(6):712-21. doi: 10.1080/10503307.2010.518636. PMID 21154029
- [Result] Teissedre F, Chabrol H. Detecting women at risk for postnatal depression using the Edinburgh Postnatal Depression Scale at 2 to 3 days postpartum. Can J Psychiatry. 2004 Jan;49(1):51-4. doi: 10.1177/070674370404900108. PMID 14763678
- [Result] Tofail F, Kabir I, Hamadani JD, Chowdhury F, Yesmin S, Mehreen F, Huda SN. Supplementation of fish-oil and soy-oil during pregnancy and psychomotor development of infants. J Health Popul Nutr. 2006 Mar;24(1):48-56. PMID 16796150
- [Result] Tofail F, Persson LA, El Arifeen S, Hamadani JD, Mehrin F, Ridout D, Ekstrom EC, Huda SN, Grantham-McGregor SM. Effects of prenatal food and micronutrient supplementation on infant development: a randomized trial from the Maternal and Infant Nutrition Interventions, Matlab (MINIMat) study. Am J Clin Nutr. 2008 Mar;87(3):704-11. doi: 10.1093/ajcn/87.3.704. PMID 18326610
- [Result] Tofail F, Hamadani JD, Mehrin F, Ridout DA, Huda SN, Grantham-McGregor SM. Psychosocial stimulation benefits development in nonanemic children but not in anemic, iron-deficient children. J Nutr. 2013 Jun;143(6):885-93. doi: 10.3945/jn.112.160473. Epub 2013 Apr 24. PMID 23616511
- [Result] Walker SP, Wachs TD, Grantham-McGregor S, Black MM, Nelson CA, Huffman SL, Baker-Henningham H, Chang SM, Hamadani JD, Lozoff B, Gardner JM, Powell CA, Rahman A, Richter L. Inequality in early childhood: risk and protective factors for early child development. Lancet. 2011 Oct 8;378(9799):1325-38. doi: 10.1016/S0140-6736(11)60555-2. Epub 2011 Sep 22. PMID 21944375
- [Result] Wolke D, Skuse D, Mathisen B. Behavioral style in failure-to-thrive infants: a preliminary communication. J Pediatr Psychol. 1990 Apr;15(2):237-54. doi: 10.1093/jpepsy/15.2.237. PMID 2374078